CLINICAL TRIAL: NCT04251338
Title: Delayed Visual Maturation: Outcome and Predictive Factors
Acronym: DVM
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S62961
Record Dates: First submitted 2019-12-31; First posted 2020-01-31 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-01

CONDITIONS: Delayed Visual Maturation
Keywords: delayed visual maturation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- delayed visual maturation: children with delayed visual maturation

SUMMARY:
The objectives of the study are to describe the developmental outcome in a population of children with delayed visual maturation.

DETAILED DESCRIPTION:
description of the developmental outcome of children with delayed visual maturation.

ELIGIBILITY:
Inclusion Criteria:

* Infants (male or female) with suboptimal/absent visual contact at the age of ≥3 months, without other known general developmental delay at the time diagnosis of delayed visual contact and without anatomic ocular abnormalities at the initial ophthalmological examination.

Exclusion Criteria:

* Children with known underlying psychomotor developmental delay or epilepsy at first ophthalmic consultation.
* Children with ophthalmic (anatomical) abnormalities that explain delayed visual maturation.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients seen in UZ Leuven between 1998 and 2016 with diagnosis of delayed visual maturation who meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
delayed visual maturation. | 1998-2016
  the prevalence of developmental problems in children with delayed visual maturation.

SECONDARY OUTCOMES:
Level of development | 1998-2016
  by questionnaire:type of education/school , problems with writing, mathematics: yes or no
Fine and gross motor skills | 1998-2016
  by questionnaire: physiotherapy needed yes or no
ophthalmological problems | 1998-2016
  by questionnaire : visual problems, wearing glasses? taped eyes?
Visual acuity | 1998-2016
  assested at the last consultation indicated in Snellen

CONTACTS AND LOCATIONS:
Overall Officials: Ingele Casteels, PhD, Principal Investigator — UZ Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No